CLINICAL TRIAL: NCT03820700
Title: The Influence of Non-pharmacological Medical Approaches Such as Hypnosis and Virtual Reality to Reduce Pain and Anxiety Before and After a Cardiovascular Surgery. A Randomized Study.
Brief Title: Using Hypnosis and Virtual Reality During Pre and Postoperative Cardiovascular Surgery.
Acronym: VRHypnICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, Responsible of the Sensation and Perception Research Group, in the GIGA CONSCIOUSNESS department, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRHICUliège
Record Dates: First submitted 2018-12-20; First posted 2019-01-29 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Thoracic Surgery; Pain, Postoperative; Anxiety; Fatigue
Keywords: Virtual Reality; Hypnosis; Intensive care units; Cardiac surgery; Anxiety; Pain; Cognition and perception; Recovery
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Fatigue; Pain | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): [Randomized] Patients in control group will receive regular nursing care but no behavioral therapy intervention.
- Hypnosis (Hypn) (Experimental): [Randomized] Patients will receive a hypnosis recorded audiotape.
  Interventions: Behavioral: Hypnosis (Hypn)
- Virtual reality (VR) (Experimental): [Randomized] Patients will see a 3D movie with a beautiful landscape.
  Interventions: Behavioral: Virtual reality (VR)
- Virtual reality hypnosis (VRH) (Experimental): [Randomized] Patients will see the same 3D film combined with a hypnotic voice.
  Interventions: Behavioral: Virtual reality hypnosis (VRH)

INTERVENTIONS:
Behavioral: Hypnosis (Hypn) — The hypnosis session will consist of a 20-minute hypnosis recording created by Marie-Elisabeth Faymonville and recorded by Anne-Sophie Nyssen, both professionals in hypnosis from University of Liège. The recording includes suggestions about relaxation, corporal sensations, respiratory techniques and visual imaginative stimuli about a beautiful landscape. With this tool, the hypnosis session is standardized for all patients and there is no need of a psychotherapist to deliver hypnosis.
  Arms: Hypnosis (Hypn)
Behavioral: Virtual reality (VR) — VR sessions. This session will consist in using a head-mounted 3D graphical display with goggles. With this tool, participants will be able to visualize a 3D immersive landscape for 20 minutes consisting of a shed near a lake at sunrise followed by a relaxing moment in the clouds. The session ends on the lake's edge.
  Arms: Virtual reality (VR)
Behavioral: Virtual reality hypnosis (VRH) — The combined tool sessions. Participants will be simultaneously subjected to the same hypnosis recording and 3D visual stimuli used in the Hypn and VR conditions.
  Arms: Virtual reality hypnosis (VRH)

SUMMARY:
Nowadays, the use of cognitive behavioral therapies has become quite common in the clinical care. Different non-pharmacological techniques, including hypnosis and virtual reality are currently used as complementary tools in the treatment of acute and chronic pain (Pourmand et al., 2017; Vanhaudenhuyse et al., 2009). A new technique called 'virtual reality hypnosis' (VRH) (Patterson et al., 2004), which encompasses a combination of both tools, is regularly used although its actual function remains unknown to this date. With the goal to improve our understanding of VRH combination effects, it is necessary to elaborate randomized and controlled research studies in order to understand their actual function in individual's perception.

100 patients who are undergoing a cardiovascular surgery at the Liège University Hospital will be randomly assigned to four conditions (control, hypnosis, VR and VRH). Each participant will receive two sessions of one of the techniques: one the day before the surgery and one other session the day after, in intensive care units.

Physiological parameters will be taken and participants will fill in a questionnaire which evaluates their level of perceived immersion, their level of anxiety, fatigue, pain and relaxation. A short interview will also be conducted to give participants the opportunity to openly describe their experience.

This study will help to expand the knowledge regarding the influence of these techniques on patient's cognition, perception and sensation .

DETAILED DESCRIPTION:
Primary outcome (anxiety) and secondary outcomes (pain, fatigue, relaxation and physiological parameters) will be investigated at four measurement times: the day before the surgery (Day -1) before the intervention (T0: baseline) and after the intervention (T1); the day after the surgery (Day+1) before the intervention (T2) and after (T3).

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing cardiac surgery
* Who have given consent for their participation.

Exclusion Criteria:

* Psychiatric antecedents
* Claustrophobia
* Acrophobia,
* Heavy hearing
* Visual impairment
* Infectious cases (example: conjunctivitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-06 (Actual); Primary Completion 2020-12-28 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Day-1 before surgery (T0 before intervention; T1 after intervention), Day+1 after surgery (T2 before intervention; T3 after the intervention)
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No anxiety = 0, maximum anxiety = 10.
Pain perception | Day-1 before surgery (T0 before intervention; T1 after intervention), Day+1 after surgery (T2 before intervention; T3 after the intervention)
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No pain = 0, maximum pain = 10.

SECONDARY OUTCOMES:
Physiological parameters | Day-1 before surgery (T0 before intervention; T1 after intervention), Day+1 after surgery (T2 before intervention; T3 after the intervention)
  Arterial pressure, heartbeat, pupil size, oxygen saturation, respiratory rates
Fatigue | Day-1 before surgery (T0 before intervention; T1 after intervention), Day+1 after surgery (T2 before intervention; T3 after the intervention)
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No fatigue = 0, maximum fatigue = 10.
Relaxation | Day-1 before surgery (T0 before intervention; T1 after intervention), Day+1 after surgery (T2 before intervention; T3 after the intervention)
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No relaxation = 0, maximum relaxation = 10.

OTHER OUTCOMES:
Participant's tendency to be absorbed and dissociated | Day-1 before surgery (T0 before the intervention)
  Dissociative Experience Scale (DES) 28-items (Beirnstein, 1986). This scale measures the dissociative experiences someone can experiment in everyday life.
Participant's opinion about the tool | Day-1 before surgery (T1 after the intervention)
  Satisfaction questionnaire created by our lab to understand if patients have a good adherence about the tool or not.
Level of absorption at the moment | Day-1 before surgery (T1 after intervention), Day+1 after surgery (T3 after the intervention)
  Absorption will be measured as the two components of hypnosis. We will measure absorption and dissociation using the Visual Analogical Scales (VAS). VAS is from 0 to 10. 0 is not absorbed and 10 is really absorbed. When responding to a VAS item, participants will be asked to specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Level of dissociation at the moment | Day-1 before surgery (T1 after intervention), Day+1 after surgery (T3 after the intervention)
  Dissociation will be measured as the two components of hypnosis. We will measure absorption and dissociation using the Visual Analogical Scales (VAS). When responding to a VAS item, participants will be asked to specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Time perception | Day-1 before surgery (T1 after intervention), Day+1 after surgery (T3 after the intervention)
  We will ask to the patient his perception of time during the session.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Vanhaudenhuyse, PhD, Study Director — CHU of Liège; Anne-Sophie Nyssen, Professor, Study Director — University of Liege
Locations (1):
- University of Liège, Liège, Province De Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rousseaux F, Dardenne N, Massion PB, Ledoux D, Bicego A, Donneau AF, Faymonville ME, Nyssen AS, Vanhaudenhuyse A. Virtual reality and hypnosis for anxiety and pain management in intensive care units: A prospective randomised trial among cardiac surgery patients. Eur J Anaesthesiol. 2022 Jan 1;39(1):58-66. doi: 10.1097/EJA.0000000000001633. PMID 34783683
- [Derived] Rousseaux F, Faymonville ME, Nyssen AS, Dardenne N, Ledoux D, Massion PB, Vanhaudenhuyse A. Can hypnosis and virtual reality reduce anxiety, pain and fatigue among patients who undergo cardiac surgery: a randomised controlled trial. Trials. 2020 Apr 15;21(1):330. doi: 10.1186/s13063-020-4222-6. PMID 32293517